CLINICAL TRIAL: NCT01212107
Title: A Phase 1 Study of LY2874455 to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy in Patients With Advanced Cancer.
Brief Title: A Phase 1 Study of LY2874455 in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13843; I4R-MC-FGAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-09-16; First posted 2010-09-30 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer; Metastatic cancer; Oncology
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Receptors, Fibroblast Growth Factor; 2-(4-(2-(5-(1-(3,5-dichloropyridin-4-yl)ethoxy)-1H-indazol-3yl)vinyl)-1H-pyrazol-1-yl)ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Part A: 2 mg FGF Receptor QD (Experimental): Part A: Dose escalation
  2 milligrams (mg) FGF receptor given orally once daily (QD) for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part A: 4 mg FGF Receptor QD (Experimental): Part A: Dose escalation
  4 mg FGF receptor given orally QD for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part A: 10 mg FGF Receptor QD (Experimental): Part A: Dose escalation
  10 mg FGF receptor given orally QD for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days).
  Interventions: Drug: FGF Receptor
- Part A: 10 mg FGF Receptor QD + Phosphate Binders (Experimental): Part A: Dose escalation
  10 mg FGF receptor + phosphate binders given QD for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor; Drug: Phosphate Binders
- Part A: 8 mg FGF Receptor BID (Experimental): Part A: Dose escalation
  8 mg of FGF receptor given orally twice a day (BID) for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part A: 10 mg FGF Receptor BID (Experimental): Part A: Dose escalation
  10 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part A: 14 mg FGF Receptor BID (Experimental): Part A: Dose escalation
  14 FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part A: 18 mg FGF Receptor BID (Experimental): Part A: Dose escalation
  18 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part A: 24 mg FGF Receptor BID (Experimental): Part A: Dose escalation
  24 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days).
  Interventions: Drug: FGF Receptor
- Part A: 18 mg FGF Receptor BID Extension (Experimental): Part A: Dose escalation
  18 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part A: 16 mg FGF Receptor BID (Experimental): Part A: Dose escalation
  16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor
- Part B: 16 mg FGF Receptor BID (Experimental): Part B: Dose determined by part a dose escalation
  16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
  If participants are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days)
  Interventions: Drug: FGF Receptor

INTERVENTIONS:
Drug: FGF Receptor — LY2874455 administered orally.
  Other Names: LY2874455
Drug: Phosphate Binders
  Arms: Part A: 10 mg FGF Receptor QD + Phosphate Binders

SUMMARY:
The study is to determine the recommended Phase 2 regimen of study drug that may be safely administered to participants with advanced and or metastatic cancer. The study consists of two parts: a dose escalation and a dose confirmation.

DETAILED DESCRIPTION:
Phase 1, first human dose study

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of cancer (solid tumors, lymphoma, or chronic lymphocytic leukemia) that is advanced and/or metastatic and for which all standard therapies have failed
* Have the presence of measurable or non-measurable disease
* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function including:

  * Hematologic: Absolute neutrophil count (ANC) equal to or greater than 1.5 x 10(9)/L platelets equal to or greater than 100 x 10(9)/L, and hemoglobin equal to or greater than 8 g/dL. Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin until 14 days after the erythrocyte transfusion
  * Hepatic: Bilirubin equal to or less than 1.5 times upper limits of normal (ULN), alanine transaminase (ALT), and aspartate transaminase (AST) equal to or less than 2.5 times ULN. If the liver has tumor involvement, AST and ALT equaling equal to or less than 5 times ULN are acceptable
  * Renal: Serum creatinine less than or equal to 1.2 times ULN or calculated creatinine clearance greater than or equal to 60 milliliters per minute using the Standard Cockcroft and Gault Creatinine Clearance Calculation
  * Calcium and phosphate less than or equal to 1.1 times ULN
* Have a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued chemotherapy and cancer-related hormonal therapy with commercially available agents for at least 21 days (6 weeks for mitomycin-C or nitrosoureas) and radiotherapy for at least 14 days prior to study enrollment and recovered from the acute effects of therapy. Hormone refractory prostate cancer participants receiving gonadotropin releasing hormone (GnRH) agonist therapy or breast cancer participants on antiestrogen therapy (for example, an aromatase inhibitor) prior to entrance on the study may have that treatment continued while they are enrolled in the study
* Females with childbearing potential must have had a negative serum pregnancy test less than or equal to 7 days prior to the first dose of study drug. Males and females with reproductive potential must agree to use 2 medically approved contraceptive methods during the trial and for 3 months following the last dose of study drug. Female participants must agree to use 2 medically acceptable methods of contraception, 1 being an oral contraceptive, dermal patch, or progestin (implantation or injection), and the other being a medically acceptable barrier method; alternatively, 2 medically acceptable barrier methods may be used. Medically acceptable barrier methods of contraception that may be used by the participant and/or his/her partner include: abstinence; diaphragm with spermicide; intrauterine device (IUD); condom together with foam, spermicide, or vaginal spermicidal suppository. Prohibited methods include the rhythm method, withdrawal, condoms alone, or diaphragm alone
* Have an estimated life expectancy of greater than or equal to 12 weeks

Exclusion Criteria:

* Have received treatment with an investigational drug, which has not received regulatory approval for any indication, within 28 days of study treatment with LY2874455
* Currently taking agents to control serum phosphate or calcium levels. This includes dietary restrictions
* Have medical conditions that, in the opinion of the investigator, would preclude participation in this study
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Participants with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic participants without history of CNS metastases is not required
* Have a history of major organ transplant (for example: heart, lungs, liver, and kidney)
* Have current acute leukemia
* Females who are pregnant or nursing
* An untreated or uncontrolled acute infection, including urinary tract infection, within 7 days of study entry
* Have Bazett's corrected QT (QTcB) greater than 470 msec (female) or greater than 450 msec (male), history of unexplained recurrent syncope, history of congenital long QT syndrome, family history of sudden death, or the presence in the screening electrocardiogram (ECG) of a conduction abnormality that in the opinion of the investigator would preclude safe participation in this study
* Have had an autologous or allogenic bone marrow transplant
* Previously treated with LY2874455

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Australia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michael M, Bang YJ, Park YS, Kang YK, Kim TM, Hamid O, Thornton D, Tate SC, Raddad E, Tie J. A Phase 1 Study of LY2874455, an Oral Selective pan-FGFR Inhibitor, in Patients with Advanced Cancer. Target Oncol. 2017 Aug;12(4):463-474. doi: 10.1007/s11523-017-0502-9. PMID 28589492

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant was defined as completer of the study after 2 cycles while a participant who discontinued was classified as a discontinuation prior to completing 2 cycles or a discontinuation after 2 cycles. Final disposition for the study is provided.
Groups:
- Part A: 2 mg FGF Receptor QD: Part A: Dose escalation
  2 milligrams (mg) FGF receptor given orally once daily (QD) for a minimum of (1) 28 day cycle.
- Part A: 4 mg FGF Receptor QD: Part A: Dose escalation
  4 mg FGF receptor given orally QD for a minimum of (1) 28 day cycle.
- Part A: 10 mg FGF Receptor QD: Part A: Dose escalation
  10 mg FGF receptor given orally QD for a minimum of (1) 28 day cycle.
- Part A: 10 mg FGF Receptor QD + Phosphate Binders: Part A: Dose escalation 10 mg FGF receptor + phosphate binders given QD for a minimum of (1) 28 day cycle.
- Part A: 8 mg FGF Receptor BID: Part A: Dose escalation
  8 mg of FGF receptor given orally twice a day (BID) for a minimum of (1) 28 day cycle.
- Part A: 10 mg FGF Receptor BID: Part A: Dose escalation 10 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
- Part A: 14 mg FGF Receptor BID: Part A: Dose escalation 14 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
- Part A: 18 mg FGF Receptor BID; Part A: 18 mg FGF Receptor BID Extension: Part A: Dose escalation
  18 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
- Part A: 24 mg FGF Receptor BID: Part A: Dose escalation
  24 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
- Part A: 16 mg FGF Receptor BID: Part A: Dose escalation 16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle
- Part B: 16 mg FGF Receptor BID (NSCLS & Gastric Cancer): Part B: Dose determined by part a dose escalation
  16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
Period: Overall Study
Arm/Group | Part A: 2 mg FGF Receptor QD | Part A: 4 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD + Phosphate Binders | Part A: 8 mg FGF Receptor BID | Part A: 10 mg FGF Receptor BID | Part A: 14 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID | Part A: 24 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID Extension | Part A: 16 mg FGF Receptor BID | Part B: 16 mg FGF Receptor BID (NSCLS & Gastric Cancer)
Started | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 58
Completed | 2 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 1 | 1 | 2 | 26
Not Completed | 1 | 1 | 3 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 32

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part A: 18 mg FGF Receptor BID: Part A: Dose escalation18 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
- Part B: 16 mg FGF Receptor BID (NSCLS & Gastric Cancer ): Part B: Dose determined by part a dose escalation 16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle
- Total: Total of all reporting groups
Arm/Group | Part A: 2 mg FGF Receptor QD | Part A: 4 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD + Phosphate Binders | Part A: 8 mg FGF Receptor BID | Part A: 10 mg FGF Receptor BID | Part A: 14 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID | Part A: 24 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID Extension | Part A: 16 mg FGF Receptor BID | Part B: 16 mg FGF Receptor BID (NSCLS & Gastric Cancer ) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 58 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (15.3) | 59.3 (14.3) | 57.8 (18.1) | 63.7 (10.5) | 65.7 (9.5) | 52.0 (11.5) | 56.7 (13.2) | 44.3 (3.8) | 55.7 (6.7) | 52.0 (24.8) | 62.7 (14.2) | 58.3 (9.5) | 57.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 19 | 30
  Male | 1 | 3 | 5 | 3 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 39 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 58 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 4 | 1 | 0 | 1 | 2 | 2 | 2 | 2 | 1 | 52 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 1 | 2 | 2 | 3 | 2 | 1 | 1 | 1 | 1 | 2 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 2 | 4 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 1 | 51 | 67
  Australia | 3 | 1 | 2 | 2 | 3 | 2 | 1 | 1 | 2 | 1 | 2 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose for Phase 2 Studies : Maximum Tolerated Dose (MTD)
Description: MTD was determined after the evaluation of Part A portion of the trial. Dose escalation proceeded at 1.3 times the preceding cohort once a Grade 3 non-laboratory toxicity or Grade 2 laboratory toxicity was noted in ≥ 1 participant until MTD was achieved. Doses up to 24 mg (48 mg/day) were evaluated in Part A. The effects at this dose and at 18 mg (36 mg/day) suggested that a reasonable number of participants might not tolerate LY2874455 for chronic administration at these dose levels because of the constellation of effects observed individually or in combination in participants at these dose levels. Therefore, the dose of 16 mg BID of LY2874455 (total dose 32 mg per day) was selected as the initial dose for Part B. Selection of the dose level was based on the tolerability of this dose and without specific toxicities identified.
Time Frame: Baseline Up to 32 Weeks
Population: All participants who received at least one dose of study drug in Part A.
Measure: Number; unit: mg
Groups:
- Part A Participants: Part A: Dose escalation
  Cohort 1: 2 milligrams (mg) FGF receptor given orally once daily (QD) for a minimum of (1) 28 day cycle.
  Cohort2: 4 mg FGF receptor given orally QD for a minimum of (1) 28 day cycle.
  Cohort3: 10 mg FGF receptor given orally QD for a minimum of (1) 28 day cycle.
  Cohort4: 10 mg FGF receptor + phosphate binders given QD for a minimum of (1) 28 day cycle.
  Cohort5: 8 mg of FGF receptor given orally twice a day (BID) for a minimum of (1) 28 day cycle.
  Cohort6: 10 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  Cohort7: 14 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  Cohort8: 18 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  Cohort9: 24 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
  Cohort10: 18 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
  Cohort11: 16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
Arm/Group | Part A Participants
Number analyzed (Participants) | 36
mg | 16

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) are events which were not present at baseline or pre-existing conditions at baseline that worsened in severity following the start of treatment. A summary of other non-serious Adverse Events (AEs), and all Serious Adverse Events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Up to 60 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: 16 mg FGF Receptor BID (NSCLS & Gastric Cancer): Part B: Dose confirmation
  16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
Arm/Group | Part A: 2 mg FGF Receptor QD | Part A: 4 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD + Phosphate Binders | Part A: 8 mg FGF Receptor BID | Part A: 10 mg FGF Receptor BID | Part A: 14 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID | Part A: 24 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID Extension | Part A: 16 mg FGF Receptor BID | Part B: 16 mg FGF Receptor BID (NSCLS & Gastric Cancer)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 58
Participants | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 58

3. Secondary Outcome: Percentage of Participants With Best Overall Response Rate (BORR) and Objective Response Rate (ORR)
Description: BORR is evaluated using response evaluation criteria in solid tumors (RECIST, version 1.1) criteria. Complete Response (CR): disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). Partial Response (PR): at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter.
  Best overall response rate = (unconfirmed CR+ unconfirmed PR) / subjects in efficacy population.
  Objective response rate = (confirmed CR+ confirmed PR) / subjects in efficacy population.
Time Frame: BORR: Baseline Up to 60 Weeks ; ORR: Baseline Up to 60 Weeks
Population: All participants who received at least one dose of study drug and who had CT Scan and progressed.
Measure: Number; unit: percentage of participants
Groups:
- Part A: 18 mg FGF Receptor BID: 18 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
- 18 mg FGF Receptor BID Extension: Part A: Dose escalation
  18 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
- Part A: 16 mg FGF Receptor BID: Part A:
  16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
Arm/Group | Part A: 2 mg FGF Receptor QD | Part A: 4 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD + Phosphate Binders | Part A: 8 mg FGF Receptor BID | Part A: 10 mg FGF Receptor BID | Part A: 14 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID | Part A: 24 mg FGF Receptor BID | 18 mg FGF Receptor BID Extension | Part A: 16 mg FGF Receptor BID | Part B: 16 mg FGF Receptor BID (NSCLS & Gastric Cancer)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 53
percentage of participants
  Best Overall Response Rate | 0 | 0 | 0 | 0 | 0 | 0 | 33.3 | 0 | 0 | 0 | 0 | 1.9
  Objective Response Rate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY2874455
Description: Maximum observed concentration during a dosing interval.
Time Frame: Part A and B: Cycle 1, Day 1, Pre-Dose, 0.5 Hr (H), 1 H, 2 H, 4H,8 H,12 H,24 H; Day 28, Pre-Dose, 0.5 H, 1 H, 2 H, 4 H, 8 H
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part B: 16 mg FGF Receptor BID (NSCLS); Part B: 16 mg FGF Receptor BID (Gastric Cancer): Part B: Dose confirmation
  16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
Arm/Group | Part A: 2 mg FGF Receptor QD | Part A: 4 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD + Phosphate Binders | Part A: 8 mg FGF Receptor BID | Part A: 10 mg FGF Receptor BID | Part A: 14 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID | Part A: 24 mg FGF Receptor BID | Part A: 16 mg FGF Receptor BID | Part B: 16 mg FGF Receptor BID (NSCLS) | Part B: 16 mg FGF Receptor BID (Gastric Cancer)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 27 | 31
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 3 | 3 | 6 | 2 | 3 | 3 | 3 | 6 | 3 | 3 | 27 | 31
  Day 1 | 6.25 (59.0) | 8.99 (27.1) | 38.4 (40.3) | 91.9 (15.1) | 27.9 (17.1) | 35.5 (52.1) | 64.9 (26.9) | 59.9 (76.3) | 107 (19.6) | 29.9 (75.6) | 63.1 (52.2) | 57.2 (61.7)
  Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 1 | 3 | 13 | 20
  Day 28 | 5.97 (66.3) | 17.1 (55.9) | 32.9 (23.0) | 36.8 (205) | 43.1 (15.2) | 63.6 (10.3) | 58.3 (12.2) | 88.6 (26.7) | 127 (NA) — n=1 only Geometric Mean available | 50.4 (167) | 79.1 (44.9) | 99.8 (38.7)

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration vs Time Curve 0 to Tau ( AUC[0-t]) of LY2874455
Description: Area under the concentration-time curve from time 0 to the end of the dosing interval (e.g., BID) calculated by a combination of linear and logarithmic trapezoidal methods (linear-up/log-down method).
Time Frame: as for outcome 4
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Groups:
- Part A:18 mg FGF Receptor BID: Part A: Dose escalation 18 mg FGF receptor given orally BID for a minimum of (1) 28 day cycle.
Arm/Group | Part A: 2 mg FGF Receptor QD | Part A: 4 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD + Phosphate Binders | Part A: 8 mg FGF Receptor BID | Part A: 10 mg FGF Receptor BID | Part A: 14 mg FGF Receptor BID | Part A:18 mg FGF Receptor BID | Part A: 24 mg FGF Receptor BID | Part A: 16 mg FGF Receptor BID | Part B: 16 mg FGF Receptor BID (NSCLS) | Part B: 16 mg FGF Receptor BID (Gastric Cancer)
Number analyzed (Participants) | 3 | 3 | 6 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 27 | 31
Hour*nanogram per milliliter (h*ng/mL)
  Day 1: number analyzed (Participants) | 3 | 3 | 6 | 2 | 3 | 3 | 3 | 6 | 3 | 3 | 27 | 31
  Day 1 | 32.7 (62.6) | 76.9 (66.7) | 224 (36.1) | 421 (18.1) | 106 (7.28) | 140 (27.3) | 301 (18.4) | 325 (85.8) | 532 (33.4) | 171 (77.2) | 291 (55.8) | 258 (66.0)
  Day 28: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 1 | 3 | 13 | 20
  Day 28 | 31.1 (92.1) | 89.7 (27.8) | 202 (13.4) | 427 (11.1) | 229 (13.2) | 301 (38.2) | 566 (9.83) | 589 (24.8) | 500 (NA) — n=1 only Geometric Mean calculable | 381 (133) | 511 (64.9) | 578 (47.3)

ADVERSE EVENTS:
Groups:
- Part A: 14 mg FGF Receptor BID: Part A: Dose escalation 14 FGF receptor given orally BID for a minimum of (1) 28 day cycle.
- Part B: 16 mg FGF Receptor BID (NSCLS and Gastric Cancer): Part B: Dose determined by part a dose escalation
  16 mg FGF Receptor given orally BID for a minimum of (1) 28 day cycle.
Arm/Group | Part A: 2 mg FGF Receptor QD | Part A: 4 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD | Part A: 10 mg FGF Receptor QD + Phosphate Binders | Part A: 8 mg FGF Receptor BID | Part A: 10 mg FGF Receptor BID | Part A: 14 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID | Part A: 24 mg FGF Receptor BID | Part A: 18 mg FGF Receptor BID Extension | Part A: 16 mg FGF Receptor BID | Part B: 16 mg FGF Receptor BID (NSCLS and Gastric Cancer)
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/6 | 0/3 | 2/3 | 1/3 | 0/3 | 2/3 | 0/3 | 1/3 | 1/3 | 18/58
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 2 mg FGF Receptor QD (N=3) | Part A: 4 mg FGF Receptor QD (N=3) | Part A: 10 mg FGF Receptor QD (N=6) | Part A: 10 mg FGF Receptor QD + Phosphate Binders (N=3) | Part A: 8 mg FGF Receptor BID (N=3) | Part A: 10 mg FGF Receptor BID (N=3) | Part A: 14 mg FGF Receptor BID (N=3) | Part A: 18 mg FGF Receptor BID (N=3) | Part A: 24 mg FGF Receptor BID (N=3) | Part A: 18 mg FGF Receptor BID Extension (N=3) | Part A: 16 mg FGF Receptor BID (N=3) | Part B: 16 mg FGF Receptor BID (NSCLS and Gastric Cancer) (N=58)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratoconjunctivitis sicca (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 2 mg FGF Receptor QD (N=3) | Part A: 4 mg FGF Receptor QD (N=3) | Part A: 10 mg FGF Receptor QD (N=6) | Part A: 10 mg FGF Receptor QD + Phosphate Binders (N=3) | Part A: 8 mg FGF Receptor BID (N=3) | Part A: 10 mg FGF Receptor BID (N=3) | Part A: 14 mg FGF Receptor BID (N=3) | Part A: 18 mg FGF Receptor BID (N=3) | Part A: 24 mg FGF Receptor BID (N=3) | Part A: 18 mg FGF Receptor BID Extension (N=3) | Part A: 16 mg FGF Receptor BID (N=3) | Part B: 16 mg FGF Receptor BID (NSCLS and Gastric Cancer) (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal lesion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 19 (38)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 16 (24)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 3 (4) | 3 (5) | 2 (2) | 3 (13) | 2 (6) | 2 (3) | 2 (3) | 45 (106)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 13 (13)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (17)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 20 (26)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 1 (4) | 1 (1) | 1 (3) | 19 (45)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 15 (24)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (3) | 2 (3) | 3 (3) | 1 (4) | 1 (2) | 1 (4) | 2 (2) | 1 (2) | 34 (47)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 1 (2) | 2 (5) | 0 (0) | 10 (19)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral fungal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Purulence (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 24 (44)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 21 (39)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 2 (12)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Calcium phosphate product increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
General physical condition abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Liver palpable subcostal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 1 (1) | 1 (2) | 2 (2) | 41 (64)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (10) | 3 (4) | 1 (1) | 2 (4) | 2 (5) | 2 (2) | 2 (5) | 46 (106)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (12)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (12)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (3) | 17 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 13 (16)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 12 (28)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days